CLINICAL TRIAL: NCT02170909
Title: Safety, Pharmacokinetics and Pharmacodynamics After Single (150 mg, 220 mg and 300 mg) and Multiple (150 mg and 220 mg q.d. and 150 mg b.i.d.) Rising Oral Doses of BIBR 1048 MS/Capsules in Healthy Male Subjects of Japanese and Caucasian Origin. (Open Label Study)
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of BIBR 1048 MS Capsule in Healthy Male Subjects of Japanese and Caucasian Origin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.29
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy

ARMS (3):
- BIBR 1048 MS low dose (Experimental)
  Interventions: Drug: BIBR 1048 MS low dose
- BIBR 1048 MS medium dose (Experimental)
  Interventions: Drug: BIBR 1048 MS medium dose
- BIBR 1048 MS high dose (Experimental)
  Interventions: Drug: BIBR 1048 MS high dose

INTERVENTIONS:
Drug: BIBR 1048 MS low dose
  Arms: BIBR 1048 MS low dose
Drug: BIBR 1048 MS medium dose
  Arms: BIBR 1048 MS medium dose
Drug: BIBR 1048 MS high dose
  Arms: BIBR 1048 MS high dose

SUMMARY:
Study to investigate and compare safety, pharmacokinetics and pharmacodynamics of BIBR 1048 MS following oral administration of single (150 mg, 220 mg and 300 mg) and multiple (150 mg and 220 mg q.d. and 150 mg b.i.d.) rising doses in healthy male subjects of Japanese and Caucasian origin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects of Japanese or Caucasian origin according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate, respiratory rate and tympanic body temperature), 12- lead ECG (electrocardiogram), clinical laboratory tests

   * 1.1 No finding deviating from normal and of clinical relevance
   * 1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥ 20 and Age ≤ 45 years
3. Body mass index (BMI) ≥ 18 and ≤ 25 kg/m2
4. Japanese subjects were from a well-defined Japanese population, both parents of Japanese origin and the subjects have Japanese passport and had lived ≤ 8 years outside Japan.
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation.

Exclusion Criteria:

1. Current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women, or an unwillingness of male subjects to use an adequate form of contraception as well as having their female partner(s) use another form of contraception (if the woman possibly become pregnant) from the time of the single dose on Day 1 until Day 22-26 (end-of study examination)
3. Current diseases of the central nervous system (such as epilepsy), or psychiatric disorders or neurological disorders
4. History of clinically significant orthostatic hypotension, clinically significant current or past fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of

   * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
   * any bleeding disorder including prolonged or habitual bleeding
   * other hematologic disease
   * cerebral bleeding (e.g. after a car accident)
   * concussions (head trauma resulting in injuring to brain) with or without loss of consciousness
7. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives, whichever is shorter, of the respective drug prior to administration or during the trial
8. Use of acetylsalicylic acid (ASA)-containing over-the-counter medications, clopidogrel or ticlopidine or dipyridamole, chronic administration of non-steroidal anti-inflammatory drugs (NSAIDs) (cyclooxygenase-2 (COX-2) inhibitors excluded), coumadin like anticoagulants, chronic use of corticosteroids, heparin and fibrinolytic agents within 14 days prior to administration or during the trial.
9. Participation in another trial with an investigational drug within three months prior to administration or during the trial
10. Smoker (> 10 cigarettes/day or > 3 cigars/day or > 3 pipes/day)
11. Inability to refrain from smoking on trial days
12. Alcohol abuse (more than 21unit/week; one unit was approximately half a pint of beer, a small glass of wine or one measure of spirits)
13. History of drug abuse
14. Blood donation (more than 100 mL within three months prior to screening administration and any blood donation from screening to end-of-study examination)
15. Excessive physical activities (within one week prior to administration or during the trial and until end-of-study examination)
16. Any laboratory value outside the reference range that was of clinical relevance
17. Inability to comply with dietary regimen of study centre
18. Known hypersensitivity to the drug or its excipients
19. History of any familial bleeding disorder
20. Thrombocytes < 150000/μL

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2004-12; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change in vital signs | Baseline and up to day 26
Change in 12-lead electrocardiogram (ECG) | Baseline and up to day 26
Change in clinical laboratory tests | Baseline and up to day 26
Occurence of adverse events | Up to day 26

SECONDARY OUTCOMES:
Area under the curve (AUC) from 0-24 hours for activated partial thromboplastin time (aPTT) | Day 1 and 12
AUC from 0-24 hours for ecarin clotting time (ECT) | Day 1 and 12
Change in thrombin time (TT) | Baseline and up to 72 hours after administration on day 1 and 12
Change in prothrombin time (PT) expressed as international normalised ratio (INR) | Baseline and up to 72 hours after administration on day 1 and 12
Maximum value of aPTT | Up to 72 hours after administration on day 1 and 12
Maximum value of ECT | Up to 72 hours after administration on day 1 and 12
Change in ECT | Baseline and up to 72 hours after administration on day 1 and 12
Change in aPTT | Baseline and up to 72 hours after administration on day 1 and 12
Cmax (maximum measured concentration of the analyte in plasma) | Up to 72 hours after administration on day 1
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | Up to 72 hours after administration on day 1
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the single dose on day 1) | Up to 72 hours after administration on day 1
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration) | Up to 72 hours after administration on day 1
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 72 hours after administration on day 1
λz (terminal rate constant in plasma) | Up to 72 hours after administration on day 1
t1/2 (terminal half-life of the analyte in plasma) | Up to 72 hours after administration on day 1
MRTpo (mean residence time of the analyte in the body after po administration) | Up to 72 hours after administration on day 1
CL/F (apparent clearance of the analyte in plasma following extravascular administration) | Up to 72 hours after administration on day 1
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular administration) | Up to 72 hours after administration on day 1
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | Up to 72 hours after administration on day 1
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | Up to 72 hours after administration on day 1
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | Up to 72 hours after administration on day 1
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 72 hours after the last dose on day 12
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | Up to 72 hours after the last dose on day 12
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 72 hours after the last dose on day 12
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 72 hours after the last dose on day 12
λz,ss (terminal rate constant in plasma at steady state) | Up to 72 hours after the last dose on day 12
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | Up to 72 hours after the last dose on day 12
MRTpo,ss (mean residence time of the analyte in the body at steady state after po administration) | Up to 72 hours after the last dose on day 12
CL/F,ss (apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration) | Up to 72 hours after the last dose on day 12
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | Up to 72 hours after the last dose on day 12
Aet1-t2,ss (amount of analyte that is eliminated in urine at steady state from the time point t1 to time point t2) | Up to 72 hours after the last dose on day 12
fet1-t2,ss (fraction of analyte eliminated in urine at steady state from time point t1 to time point t2) | Up to 72 hours after the last dose on day 12
CLR,t1-t2,ss (renal clearance of the analyte in plasma from the time point t1 until the time point t2 at steady state) | Up to 72 hours after the last dose on day 12
Accumulation ratio RA,Cmax,7 based on Cmax | Day 6 to day 15
Accumulation ratio RA,AUC,7 based on AUCτ (only for 150 mg and 220 mg q.d. groups) | Day 6 to day 15
Linearity index (LI) based on AUC (only for 150 mg and 220 mg q.d. groups) | Day 6 to day 15